CLINICAL TRIAL: NCT00002358
Title: Open-Label BV-araU Treatment of Pediatric HIV-Infected Patients With Cutaneous, Visceral, or Ocular Varicella-Zoster Viral Disease Who Have Failed or Are Intolerant of Standard Therapy
Brief Title: A Study of BV-araU in the Treatment of Varicella-Zoster Viral Disease (VZV) in HIV-Infected Children Who Have Not Had Success With or Who Cannot Take Other Treatments for VZV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 255A; AI458-903
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-10

CONDITIONS: HIV Infections; Chickenpox
Keywords: Herpes Zoster; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; sorivudine; Chickenpox
MeSH Terms: conditions — HIV Infections; Chickenpox; Herpes Zoster; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — sorivudine

INTERVENTIONS:
Drug: Sorivudine

SUMMARY:
To provide oral sorivudine ( BV-araU ) to pediatric HIV-infected patients with varicella-zoster viral disease who have failed or are intolerant of alternative therapy.

DETAILED DESCRIPTION:
Any physician qualified to treat pediatric AIDS patients may enroll patients in this study.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* Cutaneous, visceral, or ocular varicella-zoster viral infection.
* Refractory or intolerant to acyclovir or foscarnet therapy.
* Consent of parent or guardian.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Inability to take oral capsules or tolerate liquids.

Concurrent Medication:

Excluded:

* 5-flucytosine, 5-fluorouracil, high-dose prednisone, or probenecid.

Patients with the following prior condition are excluded:

History of immediate hypersensitivity to nucleoside analogues.

Prior Medication:

Excluded:

* 5-flucytosine, 5-fluorouracil, high-dose prednisone, or probenecid within 4 weeks prior to study entry.

Required:

* Prior acyclovir or foscarnet.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (1):
- Bristol - Myers Squibb Co, Wallingford, Connecticut, United States